CLINICAL TRIAL: NCT00306111
Title: Pegfilgrastim Versus Filgrastim - Intraindividual Comparison of Quantity and Quality of Mobilized Peripheral Blood Stem Cells in Patients With Non Hodgkin-lymphoma
Brief Title: Pegfilgrastim vs. Filgrastim - Comparison of Mobilized Blood Stem Cells in Patients With Non Hodgkin-lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Wolfgang Bethge, Oberarzt, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rpm_001
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2012-12

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: stem cell transplantation; stem cell mobilization; high-dose therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegfilgrastim (Experimental): Pegfilgrastim for stem cell mobilization (single arm)
  Interventions: Drug: pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim — Single dose (6mg) one day after chemotherapy
  Other Names: Neulasta(tm)

SUMMARY:
The purpose of this study is to compare the ability of pegfilgrastim vs. filgrastim to mobilize peripheral blood stem cells in patients with Non Hodgkin-lymphoma in an intraindividual study

DETAILED DESCRIPTION:
Patients with Non Hodgkin-lymphoma undergoing stem cell mobilization for planned high-dose therapy will be treated with two cycles of chemotherapy (etoposide, ifosfamide, cisplatin, epirubicin), either followed by daily administration of filgrastim (first cycle) or pegfilgrastim (once after the second cycle). The number of circulating cluster of differentiation 34+ cells, colony-forming units and primitive progenitors will be analyzed at corresponding time points. Peripheral blood stem cells will be collected after the second cycle of chemotherapy by leukapheresis. After the second cycle, high-dose therapy with peripheral blood stem cell support will be administered (the protocol will be chosen according to the diagnosis, including total body irradiation-containing regimens).

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of non-Hodgkin lymphoma
* planned high-dose therapy with autologous stem cell transplantation
* WHO performance status 0-2
* written consent

Exclusion Criteria:

* allergy against (peg)filgrastim
* life expectancy <3 months
* other malignant diseases within the last 5 years
* cardial insufficiency (>= New York Heart Association II°)
* uncontrolled infection
* pregnancy, lactation
* central nervous system lymphoma
* Karnofsky score <70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Hematopoietic recovery after autologous stem cell transplantation | 1-3 weeks after transplantation, follow up every 3 months (up to 2 years)
  Two cycles of conventional chemotherapy are given. Starting one day after the first cycle, filgrastim (5ug/kg bodyweight daily subcutaneously) is routinely administered to support neutrophil recovery. One day after the second cycle, a single dose of pegfilgrastim (6mg) is given to support neutrophil recovery and stem cell collection. Hematopoietic recovery (blood count) is monitored daily after high-dose therapy and autologous stem cell transplantation. Follow up assessments are performed 3-monthly for late graft failure

SECONDARY OUTCOMES:
Intraindividual comparison of quantity/quality of circulating stem cells | before and during 3 weeks after conventional chemotherapy
  Circulating stem cells are enumerated by flow cytometry and colony assays during filgrastim (intraindividual control) and pegfilgrastim-supported recovery from chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mohle, MD, Principal Investigator — University of Tuebingen, Dept. of Medicine 2
Locations (1):
- Dept. of Medicine 2, University of Tuebingen, Tübingen, Baden-Wurttemberg, Germany